CLINICAL TRIAL: NCT02388373
Title: A Guideline Approach to Therapy Step-down Utilising Flutiform Change and Step-down
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Napp Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR00213; 2013-005365-39 (EudraCT Number)
Record Dates: First submitted 2014-11-15; First posted 2015-03-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Seretide 250 (Active Comparator): Seretide® Evohaler® 25 microgram /50 microgram per metered dose pressurised inhalation, suspension. 25 micrograms of salmeterol (as salmeterol xinafoate) and 250 micrograms of fluticasone propionate. This is equivalent to a delivered dose (ex actuator) of 21 micrograms of salmeterol and 220 micrograms of fluticasone propionate. 2 puffs twice daily for 12 weeks Phase 1.
  Interventions: Drug: Fluticasone 250/salmeterol 25
- Flutiform 250 (Active Comparator): flutiform® 250 microgram/10 microgram per actuation pressurised inhalation, suspensions. 250 micrograms of fluticasone propionate and 10 micrograms of formoterol fumarate dihydrate. This is equivalent to a delivered dose (ex-actuator) of approximately 230 microgram of fluticasone propionate/9.0 microgram of formoterol fumarate dihydrate. 2 puffs twice daily for 12 weeks in Phase 1 and 12 weeks in Phase 2.
  Interventions: Drug: Fluticasone 250/formoterol 10
- Flutiform 125 (Active Comparator): flutiform 125 microgram/5 microgram per actuation pressurised inhalation, suspensions. 125 micrograms of fluticasone propionate and 5 micrograms of formoterol fumarate dihydrate. This is equivalent to a delivered dose (ex-actuator) of approximately 115 microgram of fluticasone propionate/4.5 microgram of formoterol fumarate dihydrate. 2 puffs twice daily for 12 weeks in Phase 2.
  Interventions: Drug: Fluticasone 125/formoterol 5

INTERVENTIONS:
Drug: Fluticasone 250/formoterol 10
  Other Names: Flutiform 250
  Arms: Flutiform 250
Drug: Fluticasone 250/salmeterol 25
  Other Names: Seretide 250 Evohaler
  Arms: Seretide 250
Drug: Fluticasone 125/formoterol 5
  Other Names: Flutiform 125
  Arms: Flutiform 125

SUMMARY:
The aim of this study is to compare two licensed asthma inhalers and to then evaluate the safety of reducing treatment when patient's asthma is in control. The inhalers used in this study are the Seretide® 250 Evohaler®, which is widely used in UK, and a recently licensed inhaler called Flutiform®. National guidelines recommend that asthma medication should be increased when patients are experiencing worsening of their asthma, and reduced when asthma is in control. However, it is likely that in daily clinical practice some patients are over-treated. It is therefore necessary to conduct more studies which demonstrate that reducing treatment dosage can be done safely.

This study has two phases. In the first phase the investigators aim to recruit 224 patients through approximately 40 clinics in the UK and Ireland. One third of these patients will be selected in random to use the high dosage Seretide® 250 Evohaler® and two thirds will use high dose Flutiform® 250 inhaler for 12 weeks. At the end of phase 1 the investigators will compare how well asthma was controlled between the two groups.

After phase 1 those patients who used Flutiform and did not have any problems with their asthma can participate in phase 2. In phase 2 half of the patients will stay on high dosage Flutiform 250 and half will be switched to the medium dosage Flutiform 125 inhaler. At the end of phase 2 the investigators will compare asthma control between the two groups.

This study will be conducted by Research in Real Life Ltd (Cambridge, UK) with partial funding from Napp Pharmaceuticals Ltd. The estimated total duration of the study is 18 months and each patient will spend a maximum of 6 months in the study.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and to comply with the study protocol.
* Current diagnosis of asthma (as evidenced by appropriate diagnostic code)
* Received Seretide® 250 Evohaler® 2 puffs twice daily for the last 6 months
* No asthma exacerbation* in last 3 months
* ≤2 exacerbations* in last 12 months
* No errors in device use after training (during baseline visit)
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after discontinuation of study drug. Acceptable methods of contraception include intrauterine device (IUD) known to have a failure rate of less than 1% per year, steroidal contraceptive (oral, implanted, transdermal, or injected), barrier method with spermicide, abstinence, and partner vasectomy.

  * Exacerbation defined as acute course of oral steroids, emergency room attendance and/or hospitalisation for asthma

Exclusion Criteria:

* Other chronic respiratory disease than asthma (e.g. Chronic Obstructive Pulmonary Disease (COPD))
* Uncontrolled asthma (GINA criteria)
* The patient has used a clinical trial investigational drug within the last year before the screening visit
* Hypersensitivity to Flutiform®, its component Formoterol or its excipients
* Pregnant subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire score (ACQ7) | 12 weeks
  At week 12 in Phase 1 and Phase 2

SECONDARY OUTCOMES:
Lung function (FEV1 and FVC) | 4 or 12 weeks
  At week 12 in Phase 1 and Phase 2 and at week 4 interim visit in Phase 2
Lung inflammation measured as level of Fractional Exhaled Nitric Oxide (FeNO) | 4 or 12 weeks
  Phase 2 only (interim visit at week 4 and final visit at week 12)
Asthma control defined by Global Initiative of Asthma (GINA) guidelines at week 12 adjusting for baseline | 4 or 12 weeks
  At week 12 in Phase 1 and Phase 2 and at week 4 interim visit in Phase 2
Visual Analog Scale (VAS) Score at week 12 adjusting for baseline | 4 or 12 weeks
  At week 12 in Phase 1 and Phase 2 and at week 4 interim visit in Phase 2
Quality of life measured with Mini Asthma Quality of Life questionnaire at week 12 adjusting for baseline | 4 or 12 weeks
  At week 12 in Phase 1 and Phase 2 and at week 4 interim visit in Phase 2
Proportion of patients with asthma control | 12 weeks
  Phase 1 and Phase 2; Asthma control defined as No exacerbations, No change in therapy, and GINA asthma control achieved
Number of adverse events | 12 weeks
  Phase 1 and Phase 2
Blood eosinophil count | Phase 2 baseline
Asthma Control Questionnaire score (ACQ7) at week 4 in Phase 2 | 4 weeks (Phase 2 interim visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Research in Real Life Ltd, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publically released as this was not covered by patient consent. Patients have consented for anonymised data to be used for future medical research by Research in Real-Life.